CLINICAL TRIAL: NCT02909595
Title: Balloon Catheter Versus Basket Catheter for Endoscopic Bile Duct Stone Extraction in Patients With Periampullary Diverticulum:a Multicenter Randomized Trial
Brief Title: Balloon Catheter vs. Basket Catheter for Endoscopic Bile Duct Stone Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Catheter001
Record Dates: First submitted 2016-09-10; First posted 2016-09-21 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-09

CONDITIONS: Biliary Calculi
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balloon catheter group (Experimental): Bile duct stones extraction was carried out with a balloon catheter.
  Interventions: Device: Balloon catheter
- Basket catheter group (Active Comparator): Bile duct stones extraction was carried out with a basket catheter.
  Interventions: Device: Basket catheter

INTERVENTIONS:
Device: Balloon catheter — Balloon stone extraction was carried out with a balloon catheter [Extractor Pro RX [M00547000, M00547010, or M00547020]; Boston Scientific,Shang hai,China). The Extractor Pro has multiple sizes (9-12, 12-15, and 15-18mm), the choice being made on the basis of the CBD diameter. It has a contrast-injection hole above the balloon for the performance of balloon occlusion cholangiography (BOC).
  Arms: Balloon catheter group
Device: Basket catheter — Basket stone extraction was performed with a basket catheter (Flower Basket V [FG-V435P or FG-V425PR]; Olympus Corp., Shang hai,China).
  Arms: Basket catheter group

SUMMARY:
Endoscopic bile duct stone (BDS) removal is a well-established treatment; however, the preference for basket or balloon catheters for extraction is operator-dependent It is reported that complete endoscopic treatment with a single catheter is more likely when choosing a balloon catheter over a basket catheter for extraction of BDSs≤10mm. However, a study comparing the two catheter types in patients with periampullary diverticulum has not been performed, and there is no strong basis on which to recommend the balloon catheter as a first-line stone removal device. The investigators therefore conducted a multicenter prospective randomized trial to compare catheter performance in patients with periampullary diverticulum.

DETAILED DESCRIPTION:
A prospective, multi-center, investigator sponsored, randomized controlled trial, 80 subjects will be randomly assigned to groups that were treated with basket or balloon catheters.

A descriptive analysis will be performed on primary endpoint, containing frequency of number and percentage of patients. A two proportion equality test will be conducted to explore whether incidence rates are different.Descriptive statistics including number (N), mean, median, standard deviation, minimum and maximum, will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age > 18 years.
2. BDSs of diameter ≤10mm, which could be extracted using a standard balloon or basket catheter without mechanical lithotripsy, and a common bile duct (CBD) diameter ≤15mm.
3. Signed inform consent form and agreed to follow-up on time

Exclusion Criteria:

1. Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent.
2. Patients involved in other study within 60 days.
3. biliary stricture
4. Billroth II or Roux-en-Y anatomy
5. Acute pancreatitis.
6. a history of previous ERCP
7. pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the rate of complete clearance of the duct in two groups. | The primary end point was the rate of complete removals of stones within 10 min.
  It has a contrast-injection hole above the balloon for the performance of balloon occlusion cholangiography (BOC). For balloon stone extraction, clearance was confirmed if no residual stones remained after the final BOC and balloon sweep. For basket stone extraction, duct clearance by the basket catheter was judged to have been completed when no filling defect was found. Complete clearance of the duct by the basket catheter was defined as no filling defect (other than air) on BOC after a balloon sweep.

SECONDARY OUTCOMES:
Secondary endpoints is the rate of adverse events such as perforation, pancreatitis,cholangitis,hyperamylasemia and bleeding. | Secondary endpoints is the rate of adverse events at 24 h after ERCP.
  If the serum amylase of patients elevation and 3 times higher than the normal values after ERCP 24 hours in patients, who also have clinical symptoms, without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc. In this condition, it will be defined PEP(post-ERCP pancreatitis). Hyperamylasemia will be defined as the serum amylase 3 times more than the upper normal values, without clinical symptoms. During the study, any unexpected medical issue will be called adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Shao Feng, MD, Principal Investigator — Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University; Wei Qi, MD, Principal Investigator — No.2 of HeFei Hospital Affiliated Anhui Medical College; YongQiang Jiang, MD, Principal Investigator — Dong fang Hospital Affiliated Anhui University Of Science & Technology
Locations (1):
- Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No